CLINICAL TRIAL: NCT00865332
Title: Psychology of Reward and Punishment: Functional and Molecular Brain Imaging and Monoaminergic Correlates
Status: Withdrawn | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Peter Herscovitch, M.D./Warren G. Magnuson Clinical Center, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080437; 08-DA-0437
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-21

CONDITIONS: Cocaine Addiction; Cocaine Abuse
Keywords: PET; fMRI; D-Amphetamine; Cocaine Addiction; Methylphenidate
MeSH Terms: conditions — Cocaine-Related Disorders

SUMMARY:
Background:

* Brain imaging studies, genetic research, and investigations of stress have provided more information about the role of dopamine in processing reward and punishment, and in vulnerability to substance dependence. Researchers are interested in learning more about how the brain responds to rewards, including drugs of abuse, and how these responses may involve genetic factors or previous stressful events.
* Researchers intend to use the drug amphetamine to increase levels of dopamine in the brain and study the effects through two kinds of scanning: functional magnetic resonance imaging (fMRI) and positron emission tomography (PET).

Objectives:

* To examine the relationship among dopamine function, brain activity, reward processing, genetic profile and exposure to stress in normal healthy adults.
* To examine the variation in these factors between normal healthy adults and individuals with current cocaine-dependence.

Eligibility:

- Individuals 18 to 45 years of age who are either current cocaine users or healthy volunteers with no history of substance abuse or dependence.

Design:

* The study will consist of an initial evaluation session and six study visits, four of which will involve fMRI scans (3 hours each) and two of which will involve PET scans (8 to 9 hours each).
* Cocaine-using participants will enter the inpatient clinical research ward at the National Institute on Drug Abuse Addiction Research Center the night before each scanning session and will be discharged the following day. Healthy volunteer subjects will not be required to stay overnight and will arrive as outpatients for the PET session. Participants will not be released until researchers have determined that participants are not experiencing significant effects of the drug.
* Initial session (1): Participants will complete questionnaires about past reactions to stressful situations, and will be trained to do thinking tasks that will be performed in fMRI visits. The tasks will be practiced in a mockup of an MRI machine.
* MRI sessions (2-5): Participants will receive either oral amphetamine or a placebo, and will perform thinking, short-term memory, and reward tasks during MRI scanning as directed by researchers.
* PET sessions (6-8): Participants will receive either oral amphetamine or a placebo, and will provide blood samples during the PET scanning sessions. Participants will have short breaks during the PET scanning sessions.

DETAILED DESCRIPTION:
Objective: This protocol will integrate functional brain imaging of reward processing, together with assessment of the response to oral dextroamphetamine (d-AMPH), monoaminergic genotyping, and evaluation of past exposure to stress, in order to examine: (1) the relationship between these factors (i.e. dopamine function, brain activity, reward processing, genetic profile and exposure to stress) in normal healthy adults; and (2) variation in these factors between normal healthy adults and individuals with current cocaine-dependence, and how this variation contributes to observed behavioral and functional differences between these populations.

Study Population: The study populations will consist of adult (18-45 years old) healthy volunteers with no history of substance abuse or dependence and a matched group of individuals with current primary cocaine-dependence.

Experimental Design and Method: After being medically cleared and giving informed consent, each participant will undergo fMRI (four sessions, on separate days) and PET scanning (two sessions, on separate days). All brain imaging sessions will take place after single-blind administration of either d-AMPH (0.43 mg/kg orally) or placebo. Functional MRI will commence after dosing and will include several measures (both cognitive and affective) designed to activate neural circuitry involved in the processing of reward and punishment. PET scanning will also take place after d-AMPH or placebo and will involve administration of the radioligand [18F] Fallypride to assess CNS dopamine function.

Outcome Measures: This study is concerned with differences in the noted factors between experimental cohorts (controls vs. cocaine-dependent adults) and conditions (baseline vs. post d-AMPH). The primary outcome measures, used to ascertain these differences, will be: (1) the percentage change in fMRI BOLD signal during performance of measures of reward processing and cognitive function; (2) alterations or differences in the binding potential of [18F]Fallypride; (3) variations in genes related to DArgic function between individuals and groups, and the contribution of this variation to other outcome measures; and (4) history of exposure to stressful events and its role in behavioral and functional outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged between 18 - 45 years;
  2. In good health, based on history and physical examination; and
  3. Right-handed (as assessed using the Edinburgh Handedness Inventory; Oldfield, 1971)

All participants in the cocaine group must meet DSM-IV criteria for cocaine dependence at the time of participation. Cocaine-dependent participants must also be positive for cocaine use in their urine toxicology screen.

EXCLUSION CRITERIA:

Potential participants for either experimental group will be excluded from participation in this study according to the following criteria:

1. Current drug use: Subjects may smoke regular cigarettes, use moderate amounts of alcohol and caffeine, or smoke an occasional marijuana cigarette. Moderate alcohol use is defined as for men, less than ten drinks and for women less than 7 drinks of liquor (1.5 oz) or the equivalent beer (12 oz) or wine (5 oz) per week. Moderate caffeine use is defined as less than 500 mg of caffeine per day, where one 5-oz serving of coffee and 2 12-oz servings of caffeinated soft drinks or tea each contain 100 mg. Occasional marijuana use is defined as less than or equal to 2 cigarettes/month. Participants may not use alcohol or marijuana for at least 24 hours prior to scanning, but will be allowed to smoke regular cigarettes according to their normal usage pattern. Participants who do not meet these guidelines for current drug use will not be allowed to participate in this study.
2. Current or Past Medication Use: Volunteers may not currently use chronic (defined as daily for more than 10/14 days in the last month) prescription or over the counter medications that might interfere with the imaging signal (PET or MRI) or which may interact adversely with any of the substances being given in this protocol. This will include, but not be limited to, anti-hypertensive, anti-allergy, and pain medications. In addition, the use of psychotropic medications, particularly antidepressants or antipsychotic medication, will be exclusionary. Past use of antidepressant medication will be evaluated on a case by case basis; however, use of MAOI's within 14 days of AMPH administration will be exclusionary due to the possibility of precipitating hypertensive crisis. Over the counter or prescription medications may be used on an occasional basis (for example, for the treatment of self-limited conditions, such as occasional headache, musculoskeletal discomfort, allergic symptoms or pain), but medications which can interact with AMPH such as Vitamin C, L-glutamine, sodium bicarbonate, and sodium phosphate will be exclusionary. In addition, current use of over-the-counter estrogen-like compounds will be exclusionary for female participants. Subjects who have previously had significant exposure to medications that act on the DA system (antipsychotics, psychostimulants) will also be excluded from the study.
3. CNS disease: History of known structural brain abnormalities (e.g. neoplasm, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g. abscess), history of head trauma (defined as documented loss of consciousness > 5 min or injury requiring hospitalization), history of seizures as an adult, sleep apnea, or tic disorder will all be exclusionary.
4. Cardiovascular, pulmonary, or systemic disease: Repeated (measured on three separate occasions) diastolic blood pressure > 90 mm Hg, or systolic blood pressure > 135 mm Hg, known arrhythmia, symptomatic or known coronary artery disease; history of endocarditis, cerebral embolism, obstructive pulmonary disease, asthma, active tuberculosis, known endocrine disease (derangements in adrenal, thyroid, bone or reproductive function), known chronic renal or hepatic dysfunction, known HIV seropositive, known current autoimmune disease involving the CNS, glaucoma, allergy to amphetamine, dextroamphetamine or known hypersensitivity to sympathomimetic amines.
5. Female participants who are currently pregnant or nursing will not be allowed to participate in this study. Female subjects will be given a serum pregnancy test a maximum of 24 hours prior to each PET session and a urine pregnancy test on the day of each fMRI session.
6. Radiation exposure: Any subject who has participated in any research studies in which he/she received a radiation exposure or has been exposed to radiation for medical or other purpose , which in combination with the present study would result in a total effective radiation exposure (from research studies) exceeding 5.0 rem in a year will be excluded.
7. Children under the age of 18 will be excluded to avoid unnecessary exposure to radiation to this population.
8. Presence in body of metallic implants or materials that could be moved by the magnet of the MRI scanner will exclude participants from this study. This will include, but not be limited to, pacemakers, surgical implants, aneurysm clips, dental braces, or bullet(s). A history of working with metal with consequent possible metal fragments in the body may also result in study exclusion.
9. Miscellaneous exclusionary criteria: Body mass greater than 300 lbs. Hematocrit < 39.0% for males or < 35.0% for females. Participants will also be excluded if veins are inaccessible.
10. Claustrophobia will also serve as an exclusion criterion.

Control Participants

In addition to those criteria outlined above, potential control participants will be excluded if they meet the following criteria:

1. Current or past psychiatric illness: DSM-IV criteria will be used (DSM-IV, APA, 1994) to determine this criterion. No subject with a current axis I diagnosis will be allowed to participate.
2. History of Drug Abuse: Control volunteers reporting either current or a significant history of illicit drug abuse (defined as single illicit substance use of more than 30 times in a lifetime for any given substance, except marijuana) will be excluded from the study.
3. Positive urine toxicology screen for either amphetamines or cocaine prior to study participation.

Cocaine-Dependent Subjects

Candidates for the cocaine-dependent group will be excluded from the study if:

1. They are actively seeking or engaged in substance abuse treatment.
2. They are dependent on other substances except nicotine or cocaine at the time of participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12-12; Study Completion 2010-12-21

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Aharon I, Etcoff N, Ariely D, Chabris CF, O'Connor E, Breiter HC. Beautiful faces have variable reward value: fMRI and behavioral evidence. Neuron. 2001 Nov 8;32(3):537-51. doi: 10.1016/s0896-6273(01)00491-3. PMID 11709163
- [Background] Angrist B, Corwin J, Bartlik B, Cooper T. Early pharmacokinetics and clinical effects of oral D-amphetamine in normal subjects. Biol Psychiatry. 1987 Nov;22(11):1357-68. doi: 10.1016/0006-3223(87)90070-9. PMID 3663788
- [Background] Arnsten AF, Goldman-Rakic PS. Noise stress impairs prefrontal cortical cognitive function in monkeys: evidence for a hyperdopaminergic mechanism. Arch Gen Psychiatry. 1998 Apr;55(4):362-8. doi: 10.1001/archpsyc.55.4.362. PMID 9554432